CLINICAL TRIAL: NCT06681662
Title: A Blinded Randomized Study of Ephedrine 0.15 Mg/kg for Reducing Onset Time of Rocuronium 0.6 Mg/kg in Elderly Patients (≥ 80 Years)
Brief Title: Ephedrine for Reducing Onset Time of Rocurinium in Elderly Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Matias Vested (Other)
Responsible Party: Sponsor-Investigator, Matias Vested, Principal Investigator, Medical Doctor, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ephedrine for rocuronium
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Ephedrine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a randomized study. Patients will be allocated randomly at a ratio of 1:1 to receive either 0.15 mg/kg ephedrine or saline (placebo). Randomization will be done at the day of operation after written informed consent is obtained. An independent investigator will allocate patients by using a computerized random number generator in REDCap. In REDCap patients also receive a number, which pseudo anonymizes data.
  The study drug is prepared in the medicine room before the operation. This is done under double control by the investigator who also performed the randomization. The study drug, either ephedrine or saline, will be prepared in a 1 mL syringe. The dose will be mixed with saline to a total of 1 mL to secure blinding.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: * The surgeon will be blinded to treatment group allocation during the induction.
  * The anesthesia personnel will be blinded to treatment group allocation during induction and intubation, but after gathering the data, they will be unblinded.
  * The investigator controlling the nerve stimulator will be blinded throughout the whole procedure.
  * Surgical personnel will be blinded to treatment group allocation during induction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ephedrine group (Active Comparator): Ephedrine 0.15 mg/kg. Dose of ephedrine is based on ideal body weight, calculated as height (cm) minus 105 for women and height (cm) minus 100 for men or actual body weight, whichever is lower.
  Interventions: Drug: Ephedrine Hydrochloride 30 mg/ml
- Saline group (Placebo Comparator): Saline 1 ml.
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Ephedrine Hydrochloride 30 mg/ml — 0.15 mg/kg during induction.
  Arms: Ephedrine group
Drug: Saline (NaCl 0,9 %) (placebo) — 1 ml during induction.
  Arms: Saline group

SUMMARY:
The aim of this study is to determine the onset time of rocuronium after administration of ephedrine 0.15 mg/kg in patients with age ≥ 80 years. The hypothesis of this study is that ephedrine 0.15 mg/kg provides a shorter onset time compared to placebo (saline).

DETAILED DESCRIPTION:
Numbers of elderly patients requiring anesthesia and surgery are increasing, and as a group, elderly patients are at high risk of postoperative complications. Aging leads to a progressive impairment of organ function and a decline in physiologic reserve and in the elderly patient population, pharmacodynamics and pharmacokinetics of medications administered during anesthesia may be influenced by the age-related reduction in cardiac output, liver function and renal function. Also, the body composition changes with age and elderly have lower total body water and an increase in body fat.

Neuromuscular blocking agents (NMBAs) are administered during anesthesia to facilitate tracheal intubation. However, in elderly patients onset time of standard doses of NMBAs are prolonged, and for 0.6 mg/kg of rocuronium it is prolonged by 50% when comparing elderly with younger adults (median 135 seconds vs 90 seconds). A prolonged onset time of rocuronium may result in prolonged time to tracheal intubation which aims to secure the patients airway and breathing during anesthesia and thereby prevents pulmonary aspiration and hypoxia. It is therefore relevant to investigate measures to reduce onset time of rocuronium in the elderly.

Ephedrine administered in younger adults undergoing general anesthesia has reduced the onset time of rocuronium 0.6 mg/kg. The mechanism behind this is speculated to be an increase in cardiac output.

It is possible to detect onset time of NMBAs with objective neuromuscular monitoring perioperatively by train-of-four (TOF) stimulation at the ulnar nerve. The effect of ephedrine on onset time of rocuronium has not been assessed in elderly patients above 80 years of age.

The possible benefit of this trial is to investigate whether ephedrine 0.15 mg/kg reduces onset time of rocuronium 0.6 mg/kg in the elderly. This may result in a shorter time to tracheal intubation and also establish better intubating conditions. The results may help to detect the optimal method for administering rocuronium to facilitate tracheal intubation in elderly patients.

The investigators hypothesize that ephedrine 0.15 mg/kg will provide a shorter onset time of rocuronium compared to placebo (saline).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 80
* Scheduled for elective operations under general anesthesia with intubation
* American Society of Anesthesiologists physical status classification (ASA) I to III
* Informed consent
* Read and understand Danish

Exclusion Criteria:

* Known allergy to rocuronium or ephedrine
* Neuromuscular disease that may interfere with neuromuscular data
* Indication for rapid sequence induction
* Daily use of beta-blocking agents
* Known cardiac arrythmia (atrial fibrillation, supraventricular or ventricular)

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Onset time of rocuronium 0.6 mg/kg defined as the time from administration of rocuronium until TOF count of 0. | Within 1 hour
  Onset time is determined by an investigator using a stop-watch.

SECONDARY OUTCOMES:
Intubating conditions assessed by The Intubation Difficulty Scale (IDS) | Within 1 hour
  Tracheal intubation will be performed when TOF count is zero. The anesthesiologist or nurse anesthetist will be interviewed after intubation by the investigator, who will note a score for each variable and the initials of the operator in the CRF. The intubating conditions will be classified with "Degree of Difficulty" according to the IDS scale, where an IDS score of 0 translates to "Easy", a score of 0 < IDS ≤ 5 translates to "Slight Difficulty" and 5 < IDS translates to "Moderate to Major Difficulty". Impossible intubation is defined by infinity (IDS = ∞ ).
Intubating conditions assessed by Fuchs-Buder scale | Within 1 hour
  Tracheal intubation will be performed when TOF count is zero. The anesthesiologist or nurse anesthetist will be interviewed after intubation by the investigator, who will note a score for each variable and the initials of the operator in the CRF. All variables will be assessed as either excellent, good or poor. The intubating conditions will be classified as excellent if all qualities are excellent, good if all qualities are either excellent or good and poor if the presence of a single quality listed as poor.
Occurrence of new cardiac arrythmia during induction of anaesthesia (<15 minutes after administration of ephedrine or saline) | Within 15 minutes
Change in mean arterial blood pressure from before induction to immediately after intubation | Within 1 hour
Time to TOF 0.9 | Within 4 hours

OTHER OUTCOMES:
Occurrence of hoarseness and sore throat 24 and 72 hours postoperatively | Within 72 hours
  After 24 hours patients are asked about hoarseness and sore throat. The patients who experience either or both will be called 3 days postoperatively again. These two variables are assessed using a numeric ranking scale.

CONTACTS AND LOCATIONS:
Overall Officials: Matias Vested, Study Chair — Rigshospitalet, University of Copenhagen
Locations (2):
- Denmark (2):
  - Department of Anaesthesiology, Pain and Respiratory Support, Rigshospitalet Glostrup, Copenhagen
  - Department of Anesthesia, Centre of Head and Orthopedics, 6013 Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No